CLINICAL TRIAL: NCT06904170
Title: An Integrated Phase II/III Randomized Study Comparing Durvalumab and Tremelimumab +/- Hepatic ArteriaL Infusion Chemotherapy With GEMOX in Hepatocellular Carcinoma With High Tumor burdEn
Brief Title: Durvalumab and Tremelimumab With or Without Hepatic Arterial Infusion of Chemotherapy in Hepatocellular Carcinoma
Acronym: ALICE
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-GIG-2406; 2024-514912-28-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-09; First posted 2025-04-01 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: High tumor burden, HAIC, GEMOX, HCC,
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Durvalumab + Tremelimumab (single dose), combined with Hepatic Arterial Infusion Chemotherapy (HAIC) of gemcitabine + oxaliplatin (GEMOX regimen)
  Interventions: Drug: Durvalumab Plus Tremelimumab; Drug: HAIC (GEMOX)
- Arm B (Active Comparator): Durvalumab + Tremelimumab (single dose)
  Interventions: Drug: Durvalumab Plus Tremelimumab

INTERVENTIONS:
Drug: Durvalumab Plus Tremelimumab — Systemic infusion of :
  Tremelimumab 300 mg, single dose at Cycle 1 Durvalumab 1500 mg at Cycle 1 then every 4 weeks until disease progression or unacceptable toxicity.
  Durvalumab and Tremelimumab will be delivered during a single angiography. Implantable catheter is also allowed.
  Durvalumab infusion will start 1 hour after the end of the tremelimumab infusion.
Drug: HAIC (GEMOX) — Hepatic Arterial Infusion of Chemotherapy (HAIC) :
  Gemcitabine 1000 mg/m² over 30 minutes, followed by Oxaliplatin 100 mg/m² over 2 hours. Administered every 2 weeks for 4 cycles. When a Durvalumab cycle match with an HAIC infusion, HAIC will be delivered on the same day.
  Arms: Arm A

SUMMARY:
Liver cancer is a highly lethal malignancy and has become increasingly important in western countries. The management of liver cancer is complex. In advanced disease, two combinations of immunotherapies are recommanded as first line (atezolizumab-bevacizumab or durvalumab-tremelimumab). Results in patients with high tumor burden (Portal vein thrombosis Vp3 or Vp4, or tumoral liver involvement >50%) are less impressive. Innovative combinations are necessary to improve the outcome of patients.

Recently, control trials conducted in Asia highlighted the benefit of hepatic arterial infusion chemotherapy, especially in patients with high tumor burden. Studies including a limited number of patients shown that the combination seems feasible.

ALICE is a randomized multicentric Phase II/Phase III trial conducted in French medical centers, evaluating the efficacy and safety of durvalumab+tremelimumab with or without Hepatic Arterial Infusion Chemotherapy of the GEMOX regimen (gemcitabine + oxaliplatin), in patients with high tumor burden.

Oxaliplatin induce immunogenic cell death, and gemcitabin deplete regulatory immune cells. The GEMOX regimen thus has the potential for a synergic effect with immunotherapy in HCC.

The trial will provide an innovative treatment to patients with no alternative for locoregional treatment, and with limited results with actual systemic treatments. It will also be the first trial of Hepatic Arterial infusion for such patients in the western population.

DETAILED DESCRIPTION:
The ALICE study will randomize 196 patients in about 20 sites in France, according to a ratio 1:1, and in 2 steps :

* 90 Patients will first be included in the initial Phase II study, and compared in terms of ORR.
* 106 additional patients with be included for the Phase III, and the total population will be analyzed in terms of Overall Survival.

A safety run-in phase will be planned for the first 12 patients in the experimental arm, to assess the tolerance of the treatment combination. An independent Study Monitoring Board (DSMB), with expertise and experience in the pathology, and without direct involvement in the conduct of the study, will be set up specifically to ensure optimal safety monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old,
* Patient presenting with hepatocellular carcinoma (HCC), diagnosed either by histological or radiological criteria as described by EASL criteria, if no biopsy could be performed safely.
* High-tumor burden, defined as at least one of the three criteria: (i) Vp4 PVTT, (ii) Vp3 PVTT with bilobar tumoral involvement and/or (iii) liver involvement >50% (as assessed by the investigator). Extra-hepatic spread is allowed.
* Child-Pugh A liver function
* Performance status Eastern Cooperative Oncology Group (ECOG) 0 to 1
* Must have a life expectancy of at least 12 weeks
* Body weight >30 kg
* At least 1 lesion, not previously irradiated, that qualifies as a RECIST 1.1 target lesion (TL) at baseline. Tumor assessment by computed tomography (CT) scan or magnetic resonance imaging (MRI) must be performed within 28 days prior to randomization
* Adequate organ and marrow function as indicated by the following laboratory values

  1. Haemoglobin ≥ 7.5 g/dL. Participants with 7.5 g/dL < haemoglobin < 9.0 g/dL having active or chronic bleeding to be excluded,
  2. Platelet count ≥75 × 109/L,
  3. Absolute neutrophil count (ANC ≥1.0 × 109 /L)
  4. creatinine clearance > 40 mL/min (according to Cockcroft or MDRD formula)
  5. AST (SGOT)/ALT (SGPT) ≤5x ULN
  6. Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN).
  7. International normalised ratio (INR) < 2.3
* Women of childbearing potential must be willing to use a highly effective method of birth control for the duration of the study, and ≥90 days after the last dose of study drug, and have a negative urine or serum pregnancy test ≤7 days of first dose of study drug. In case of a urine pregnancy test, it must be a highly sensitive urine pregnancy test.
* Non-sterile males must be willing to use a highly effective method of birth control for the duration of the study and for ≥90 days after the last dose of study drug. A sterile male is defined as one for whom azoospermia has been previously demonstrated in a semen sample examination as definitive evidence of infertility. Males with known "low sperm counts" (consistent with "sub-fertility") are not to be considered sterile for purposes of this study.
* Men and women patients must consent to not donate or bank sperm or ova during treatment and for 180 days after treatment stop
* Patients must have provided consent for the study by signing and dating a written informed consent form prior to any study specific procedures, sampling, or analyses. When the patient is physically unable to give their written consent, a trusted person of their choice, independent from the investigator or the sponsor, can confirm in writing the patient's consent
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
* Patient affiliated to a social security regimen

Exclusion Criteria:

* Previous systemic treatment (either immunotherapy, anti-angiogenics, chemotherapy, or any combination thereof)
* Previous treatment with hepatic arterial infusion of chemotherapy
* Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.
* History of hepatic encephalopathy within the past 6 months or requirement for medications to prevent or control encephalopathy (eg, no lactulose, rifaximin, etc if used for purposes of hepatic encephalopathy).
* Active or prior documented gastrointestinal bleeding (GI; eg, esophageal varices or ulcer bleeding) within the past 6 months. Note: For participants with a history of GI bleeding greater than 6 months or assessed as high risk for esophageal varices by the investigator, including main trunk portal vein thrombosis, a recent endoscopy within 3 months of enrolment and adequate endoscopic therapy according to institutional standards is required.
* Any unresolved toxicity NCI CTCAE grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

  1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
  2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Study Physician.
* Any concurrent chemotherapy, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

  1. Patients with vitiligo or alopecia
  2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  3. Any chronic skin condition that does not require systemic therapy
  4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician
  5. Patients with celiac disease controlled by diet alone
* History of interstitial lung disease, non-infectious pneumonitis or uncontrolled diseases including pulmonary fibrosis, acute lung diseases
* History of leptomeningeal carcinomatosis
* Known active hepatitis infection, positive hepatitis C virus (HCV) antibody, hepatitis B virus (HBV) surface antigen (HBsAg) or HBV core antibody (anti-HBc), at screening. Participants with a past or resolved HBV infection (defined as the presence of anti HBc and absence of HBsAg) are eligible. Participants positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Known to have been tested positive for human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies) or active tuberculosis infection (clinical evaluation that may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice).
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea
* Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart)
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* Receipt of live attenuated vaccine within 30 days prior to the first dose of study drug
* History of allogenic organ transplantation, or patient with intent for transplantation
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of study drug. Note: Local surgery of isolated lesions for palliative intent is acceptable
* Prior malignancy active within the previous 5 years of inclusion except for locally curable cancers considered cured or successfully resected, such as basal or squamous cell skin cancers, superficial bladder cancer, or gastric cancers, or carcinoma in situ of the prostate, cervix, or breast carcinomas. Any oncological concomitant treatment is not allowed during the treatment period.
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy or180 days after the last dose of durvalumab and tremelimumab combination therapy.
* Participation in another therapeutic trial within the 30 days prior to study inclusion
* Prior randomisation or treatment in a previous durvalumab and/or tremelimumab clinical study regardless of treatment arm assignment.
* Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* Patients deprived of their liberty or under protective custody or guardianship
* Patients unable to adhere to the protocol for geographical, social, or psychological reasons or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2029-09-14 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Phase II : Objective Response Rate according to RECIST 1.1 | From date of randomization until the date of first documented progression, and up to 6 months after the inclusion of the last patient
  The proportion of patients with Complete Response or Partial Response according to RECIST 1.1
Phase III : Overall Survival | From date of randomization to the date of death, up to 18 months after the randomization of the last patient
  The time between Randomisation and death from any cause

SECONDARY OUTCOMES:
Safety of the combination of immune therapy and HAIC | From the first study treatment administration to 30 days after the last administration of study treatment
  Will be assessed :
  * the frequency of limiting toxicities (LT) occuring during the combination phase (the first 12 weeks). LT are defined as any toxicity related to the experimental drug, that leads to definitive treatment discontinuation.
  * the frequency and severity of treatment-related adverse events as per NCI-CTCA v5.0
Progression-Free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever occurs first, up to 18 months after the inclusion of the last patient
  Defined as the delay between the date of randomization and the date of the first progression or death from any cause. Progression will be assessed via RECIST 1.1 and mRECIST.
Phase II : Overall Survival | From date of randomization to the date of death, up to 18 months after the randomization of the last patient
  Defined as the delay between randomization and death from any cause.
Phase III : Objective Response Rate | From date of randomization until the date of first documented progression, and up to 6 months after the inclusion of the last patient
  Defined as the proportion of patients with Complete Response or Partial Response according to RECIST 1.1
Health-Related Quality of Life (HRQoL) measured by the EORTC QLQ-C30 questionnaire | From date of randomization and until the date of first documented progression, up to 18 months after the inclusion of the last patient
  Quality of life will be assessed with questionnaire EORTC QLQ-C30, at baseline and every 2 months until disease progression or study termination
Health-Related Quality of Life (HRQoL) measured by the EORTC HCC-18 questionnaire | From date of randomization and until the date of first documented progression, up to 18 months after the inclusion of the last patient
  Quality of life will be assessed with questionnaire EORTC HCC-18, at baseline and every 2 months until disease progression or study termination

CONTACTS AND LOCATIONS:
Overall Officials: Julien EDELINE, Professor, Principal Investigator — Centre Eugène Marquis; Laure Monard, Study Director — UNICANCER
Locations (11):
- France (11):
  - CHU de Bordeaux, Bordeaux
  - AP-HP Hôpital Beaujon, Clichy
  - Centre Georges Francois Leclerc, Dijon
  - Hôpital Saint Joseph, Marseille
  - CHU de Montpellier, Montpellier
  - CHU Hôtel-Dieu, Nantes
  - AP-HP Hôpital Cochin, Paris
  - CHU de Poitiers, Poitiers
  - Centre Eugene Marquis, Rennes
  - CHRU de Strasbourg, Strasbourg
  - CHU de Rangueil, Toulouse

IPD SHARING:
Plan to Share IPD: No